CLINICAL TRIAL: NCT07356375
Title: PROMISE: Evaluation of Patient-Reported Outcomes and Adherence After Transition From Inhaled Iloprost to Oral Selexipag in Pulmonary Arterial Hypertension
Brief Title: Patient-Reported Outcomes and Adherence After Transition From Inhaled Iloprost to Oral Selexipag in Pulmonary Arterial Hypertension
Acronym: PROMISE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Caio Júlio César dos Santos Fernandes, MD, University of Sao Paulo General Hospital
Other Study IDs: SGP 27905
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: Pulmonary Arterial Hypertension; Prostacyclin Pathway; Patient-Reported Outcomes; Quality of Life; Treatment Adherence; Real-World Evidence; Iloprost; Selexipag; Observational Study
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Treatment Adherence and Compliance | interventions — selexipag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Iloprost to Selexipag Transition: Adult patients with pulmonary arterial hypertension receiving inhaled iloprost whose treating physician decides, as part of routine clinical care, to transition treatment to oral selexipag. Patients are followed prospectively to assess changes in patient-reported outcomes, treatment satisfaction, and adherence before and after the transition. All treatment decisions are made by the treating physician, and no study-related intervention is performed.
  Interventions: Drug: Selexipag

INTERVENTIONS:
Drug: Selexipag — Exposure to oral selexipag following transition from inhaled iloprost as part of routine clinical care in adults with pulmonary arterial hypertension. The decision to initiate, titrate, or discontinue selexipag is made exclusively by the treating physician, independent of study participation. No study-mandated intervention or treatment assignment is performed. The study observes patient-reported outcomes, treatment satisfaction, and adherence associated with this treatment transition.
  Other Names: Oral selexipag; IP receptor agonist

SUMMARY:
Pulmonary arterial hypertension (PAH) is a rare and serious condition that affects the blood vessels of the lungs and can significantly limit daily activities and quality of life. Some patients with PAH use inhaled iloprost, a medication that requires several inhalations per day, which can be difficult to maintain over time. Oral selexipag is an alternative treatment that may reduce treatment burden and improve adherence.

The PROMISE study aims to evaluate how switching from inhaled iloprost to oral selexipag affects patients' quality of life, satisfaction with treatment, and adherence in real-world clinical practice. Patient-reported outcome questionnaires will be used to understand patients' perceptions of symptoms, daily functioning, and overall improvement after the transition.

Adult patients with PAH who are receiving inhaled iloprost and whose physicians decide to switch treatment to oral selexipag will be followed over time. A comparison group of patients who continue using inhaled iloprost will also be observed. The study does not involve any experimental treatment or changes to routine clinical care. All medications are prescribed as part of standard medical practice.

The results of this study may help improve understanding of the patient experience during treatment transitions in PAH and support more patient-centered treatment decisions.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a progressive and life-threatening disease that requires long-term treatment with targeted therapies. Medications acting on the prostacyclin pathway are an important component of PAH management. Inhaled iloprost has demonstrated clinical and hemodynamic benefits but requires multiple daily inhalations, which may increase treatment burden and negatively affect adherence and daily functioning. Oral selexipag, a selective IP receptor agonist administered twice daily, offers a less complex dosing regimen and may improve treatment persistence and patient experience.

In Brazil, the incorporation of oral selexipag into national treatment guidelines has led to an increasing number of patients transitioning from inhaled iloprost to oral therapy as part of routine clinical care. However, data on patient-reported outcomes, satisfaction, and real-world adherence following this transition are limited, particularly in Latin American populations.

The PROMISE study is a prospective, observational, single-center study designed to assess the patient experience associated with the transition from inhaled iloprost to oral selexipag in adults with PAH. The study focuses on changes in health-related quality of life, treatment satisfaction, global perception of improvement, and objective and self-reported measures of adherence over time. A comparison group of patients who continue treatment with inhaled iloprost will be followed in parallel to provide contextual interpretation of observed changes.

All treatment decisions, including initiation, continuation, titration, or discontinuation of medications, are made exclusively by the treating physician according to standard clinical practice. Participation in the study does not influence therapeutic choices, and no additional interventions beyond routine care are performed. Data collection consists of validated patient-reported outcome measures, structured questionnaires, and review of clinical information obtained during usual follow-up visits.

By capturing patient-centered outcomes in a real-world setting, the PROMISE study aims to improve understanding of the impact of treatment transitions on daily life and adherence in PAH, supporting more informed, patient-focused management strategies.

ELIGIBILITY:
Inclusion Criteria

Adults aged 18 years or older.

Confirmed diagnosis of pulmonary arterial hypertension (PAH, Group 1) by right heart catheterization.

Current treatment with inhaled iloprost as part of routine clinical care.

Clinical decision by the treating physician to transition from inhaled iloprost to oral selexipag.

Ability to understand and complete patient-reported outcome questionnaires.

Provision of written informed consent.

Exclusion Criteria

Significant cognitive impairment or sensory deficits that prevent completion of study questionnaires.

Unstable or decompensated comorbid conditions that may interfere with treatment adherence or study participation.

Refusal or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with a confirmed diagnosis of pulmonary arterial hypertension (PAH, Group 1) who are receiving inhaled iloprost as part of routine clinical care at a specialized referral center. Eligible patients are those for whom the treating physician has decided, based on clinical judgment, to transition therapy from inhaled iloprost to oral selexipag. Participants are followed prospectively to assess patient-reported outcomes, treatment satisfaction, adherence, and safety associated with this treatment transition. All clinical decisions are made independently of study participation, and no study-mandated interventions are performed.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life (EMPHASIS-10) | From baseline (prior to transition) to 16-24 weeks of follow-up
  Change in health-related quality of life assessed by the EMPHASIS-10 questionnaire, measured as the difference in total score between baseline (prior to transition from inhaled iloprost to oral selexipag) and follow-up. Lower scores indicate better quality of life. The primary outcome evaluates within-patient change after the treatment transition in routine clinical practice.

SECONDARY OUTCOMES:
Change in Treatment Satisfaction (TSQM-9) | From baseline (prior to transition) to 3-4 weeks and 16-24 weeks after transition
  Change in treatment satisfaction assessed using the Treatment Satisfaction Questionnaire for Medication (TSQM-9), measured before the transition from inhaled iloprost and after transition to oral selexipag. The TSQM-9 evaluates effectiveness, convenience, and global satisfaction domains, allowing within-patient comparison of treatment satisfaction before and after the switch.
Patient Global Impression of Change (PGIC) | 3-4 weeks and 16-24 weeks after transition
  Patient-reported global impression of change assessed using the PGIC scale, reflecting the patient's overall perception of improvement or worsening following the transition from inhaled iloprost to oral selexipag, and its correlation with changes in patient-reported outcomes.
Objective Adherence to Selexipag | From transition to 16-24 weeks of follow-up
  Objective treatment adherence assessed by the percentage of days with twice-daily selexipag use, treatment interruptions, and the highest titrated dose achieved during follow-up, as documented in routine clinical practice.
Perceived Treatment Burden | From baseline (prior to transition) to 16-24 weeks after transition
  Perceived treatment burden evaluated before the transition, based on the number of daily inhalations with iloprost, and after the transition, based on patient-reported convenience of the oral selexipag regimen.
Adverse Events and Health Care Utilization | From transition to 16-24 weeks of follow-up
  Occurrence of adverse events and health care utilization, including hospitalizations and unplanned outpatient visits, recorded during routine clinical follow-up after transition to oral selexipag.
Responder Status Based on EMPHASIS-10 | From baseline to 16-24 weeks of follow-up
  Proportion of patients achieving a clinically meaningful improvement in health-related quality of life, defined as a decrease of at least 6 points (minimal clinically important difference) in the EMPHASIS-10 score between baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Caio Fernandes, MD, Principal Investigator — UNIVERSIDADE SAO PAULO

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Simonneau G, Montani D, Celermajer DS, Denton CP, Gatzoulis MA, Krowka M, et al. Haemodynamic definitions and updated clinical classification of pulmonary hypertension. Eur Respir J. janeiro de 2019;53(1):1801913. 2. Humbert M, Sitbon O, Simonneau G. Treatment of Pulmonary Arterial Hypertension. N Engl J Med. 30 de setembro de 2004;351(14):1425-36. 3. Calderaro D, Alves Junior JL, Fernandes CJCDS, Souza R. Pulmonary Hypertension in General Cardiology Practice. Arq Bras Cardiol [Internet]. 2019 [citado 24 de agosto de 2024]; Disponível em: https://www.scielo.br/scielo.php?pid=S0066-782X2019000900419&script=sci_arttext 4. Yoo HHB. Lesões Plexiformes na Hipertensão Arterial Pulmonar: Estamos Ficando mais Próximos do Manejo com mais Paciência e Rigor? Arq Bras Cardiol. 18 de setembro de 2020;115(3):491-2. 5. D'Alonzo GE, Barst RJ, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, et al. Survival in patients with primary pulmonary hypertension. Results from a national prospective registry. Ann Intern Med. 1o de setembro de 1991;115(5):343-9. 6. Barst RJ, Rubin LJ, Long WA, McGoon MD, Rich S, Badesch DB, et al. A comparison of continuous intravenous epoprostenol (prostacyclin) with conventional therapy for primary pulmonary hypertension. N Engl J Med. 1o de fevereiro de 1996;334(5):296-301. 7. Galiè N, Ghofrani HA, Torbicki A, Barst RJ, Rubin LJ, Badesch D, et al. Sildenafil citrate therapy for pulmonary arterial hypertension. N Engl J Med. 17 de novembro de 2005;353(20):2148-57. 8. Rubin LJ, Badesch DB, Barst RJ, Galiè N, Black CM, Keogh A, et al. Bosentan Therapy for Pulmonary Arterial Hypertension. N Engl J Med. 21 de março de 2002;346(12):896-903. 9. Hoeper MM, Badesch DB, Ghofrani HA, Gibbs JSR, Gomberg-Maitland M, McLaughlin VV, et al. Phase 3 Trial of Sotatercept for Treatment of Pulmonary Arterial Hypertension. N Engl J Med. 20 de abril de 2023;388(16):1478-90. 10. Mitchell JA, Ahmetaj-Shala B, Kirkby NS, Wright WR, Mackenzie LS, Reed DM, et al. Role of pr